CLINICAL TRIAL: NCT00376116
Title: Home CARE - Home Monitoring in CArdiac REsynchronisation Therapy
Brief Title: Home Monitoring in Cardiac Resynchronisation Therapy
Acronym: HomeCARE
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Other Study IDs: TA056
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2008-11-17 (Estimated); Status verified 2008-11

CONDITIONS: Heart Failure, Congestive
Keywords: Implantable cardioverter-defibrillator; Pacemaker; Cardiac resynchronisation therapy; Heart failure; Predictor; Mortality; Rehospitalization; Telemedicine; Home Monitoring
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy; Defibrillators, Implantable

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Cardiac resynchronisation therapy
Device: Implantable cardioverter-defibrillator

SUMMARY:
In spite of success in the management of heart failure, repetitive rehospitalisation and high mortality rate remain a serious problem. Recent studies, especially the COMPANION trial, have demonstrated that cardiac resynchronisation therapy (CRT) reduces mortality and rehospitalisation in heart failure patients. There is also evidence that telemonitoring of heart failure patients potentially reduces both mortality and morbidity. Recently, a Home Monitoring (HM) function has been integrated into BIOTRONIK CRT-defibrillators and CRT-pacemakers with a view of harnessing the powerful combination of CRT with close remote monitoring of heart failure patients. It is possible now to transmit predefined parameters on a daily basis from the implanted devices to a web-based platform accessible by patients' physicians. Our study evaluates clinical usefulness of Biotronik HM function in CRT-defibrillators and CRT-pacemakers.

DETAILED DESCRIPTION:
Clinical investigations identified potential predictors for mortality and rehospitalisation events in heart failure patients. A selection of these predictors primarily composes the "Heart Failure Monitor" (HFM), which is implemented in Biotronik implantable cardioverter defibrillators (ICDs) capable of delivering cardiac resynchronisation therapy (CRT) as well as in CRT-pacemakers. HFM and other parameters are transmitted to the attending physician via Home Monitoring (HM) function integrated in the implanted devices. In the future, a HFM with high predictive power may play an important role as part of a strategy of delivering effective health care for heart failure patients with an indication for CRT.

Our included patients implanted with CRT devices STRATOS LV-T (CRT-pacemaker), KRONOS LV-T, or Lumax HF-T (CRT-ICD). Pre-discharge protocol comprised standard device follow-up, activation of the HM-function, and assessment of complications and cardiovascular events. At follow-up controls 1, 3, 6, 9, and 12 months after implantation, standard device follow-up was performed and complications and cardiovascular events were assessed.

At enrollment, 6 and 12 months postoperative and in case of a rehospitalisation, the following parameters are documented:

* Echocardiographic parameters
* Quality of Life (Minnesota)
* ECG-parameters, NYHA-classification
* Blood pressure, body weight
* BNP / NT-pro BNP (optional)
* 6 minute walk test (optional)

At 1, 3 and 9 months postoperative:

* ECG-parameters, NYHA-classification
* Blood pressure, body weight
* BNP / NT-pro BNP (optional)
* 6 minute walk test (optional)

Further documentation:

* Change of drug treatment
* Any cardiovascular event and therapeutic intervention
* Heart failure related symptoms by means of patient diary

ELIGIBILITY:
Inclusion Criteria:

* Written patient informed consent
* Indication for CRT (biventricular or bifocal)
* Sufficient GSM-network coverage in the patient's area
* Stable residence during follow-up (anticipated)
* at least 1 documented hospitalisation due to heart failure within 12 months before enrolment

Exclusion Criteria:

* Permanent atrial fibrillation
* Myocardial infarction or instable Angina Pectoris within the last 3 months
* Planned cardiac interventions within the next 3 months (e.g. PTCA, CABG, HTX)
* Acute myocarditis
* Life expectancy under 6 months
* Pregnant or breast-feeding woman
* Participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2005-03; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of (single or combined) HFM-parameters (onset of arrhythmias, duration of physical activity, mean heart rate at rest and over 24h, %CRT, lead impedance)
Predictive power of HFM-parameters regarding cardiovascular-based death or rehospitalisation (overnight stay)

SECONDARY OUTCOMES:
Effectiveness of HM (within sub-study)
Correlation of HM-values with the clinical status
Evaluation of the predictive power of HM parameters not implemented in the HFM and of parameters not transmitted by HM (diagnostic memory of device)
Sensitivity of HM-parameter regarding change of drug therapy
Incidence and reasons for HM-based interventions

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sack, Associate Prof. Dr., Principal Investigator — Division of Cardiology, University of Essen, Germany; Vincent Paul, MD, Principal Investigator — Cardiology Department, St. Peter's Hospital, Chertsey Surrey, United Kingdom
Locations (82):
- Austria (2):
  - LKH-Universitätsklinikum Graz, Graz
  - Medizinische Universität Wien, Vienna
- Czechia (3):
  - Fakultni nemocnice u Svety Anny, Brno
  - IKEM, Prague
  - Petr Neuzil M.D., Ph.D., Prague
- France (9):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital Cardiologique du Haut Lévêque, Bordeaux
  - CHU de Lyon - Hôpital Louis Pradel, Lyon
  - Groupe Hospitalier de la Timone, Marseille
  - CHRU Hôpital de Villeneuve, Cardiologie A, Montpellier
  - CHRU Hôpital de Villeneuve, Cardiologie B, Montpellier
  - Centre Hospitalier, Pau
  - Hôpital haut Lévêque, Pessac
  - CHU des Rennes, Rennes
- Germany (51):
  - Universitätsklinik der RWTH Aachen, Aachen
  - Helios Klinikum Aue GmbH, Aue
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Krankenhaus Bassum, Bassum
  - Evangelisches Krankenhaus, Bergisch Gladbach
  - Gemeinschaftpraxis für Kardiologie und Angiologie, Bergisch Gladbach
  - Universitätsklinikum Charité, Berlin
  - Ambulantes Herzzentrum, Berlin
  - Franz-Volhard-Klinik, Berlin
  - Campus Virchow Klinikum, Charité, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Städtische Kliniken Bielefeld gGmbH, Bielefeld
  - Berufsgenossenschaftliche Kliniken Bergmannsheil, Bochum
  - Praxisgemeinschaft, Braunschweig
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Zentralkrankenhaus Links der Weser, Bremen
  - Kardiologische Gemeinschaftspraxis, Chemnitz
  - Klinikum Coburg, Coburg
  - Herzzentrum Coswig, Coswig
  - Carl-Thiem-Klinikum, Cottbus
  - Cardiac Research GmbH, Dortmund
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Praxiszentrum Herzkreislauf, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Elisabeth Krankenhaus Essen, Essen
  - Klinikum Frankfurt/Oder GmbH, Frankfurt (Oder)
  - Ernst-Moritz-Arndt Universität Greifswald, Greifswald
  - Allgemeines Krankenhaus Altona, Hamburg
  - Kardiologische Gemeinschaftspraxis, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Praxis Dr. med. Natour, Heidelberg
  - Medizinische Universitätsklinik Homburg/Saar, Homburg/Saar
  - Klinikum Hoyerswerda, Hoyerswerda
  - Gemeinschaftspraxis Dr. Kroll/Dr. Rebeski, Kiel
  - Herzzentrum Konstanz GmbH, Konstanz
  - PD Dr. Christoph Karle, Künzelsau
  - Städtisches Klinikum St. Georg, Leipzig
  - Herzzentrum Leipzig GmbH, Leipzig
  - Märkische Kliniken GmbH, Lüdenscheid
  - Klinikum Johannes-Gutenberg-Universität, Mainz
  - Praxis Dr. Patrizia Kindler, Meiningen
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Stiftsklinik Augustinum, München
  - Ruppiner Klinikum GmbH, Neuruppin
  - Klinikum Pirna GmbH, Pirna
  - St. Adolf-Stift, Reinbek
  - St. Elisabeth Klinik, Saarlouis
  - Kardiologische Gemeinschaftspraxis Dr. Hoh u. Dr. Tamm, Wittenberg/Lutherstadt
  - Universitätsklinikum Würzburg, Würzburg
- Israel (5):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, ICCU, Ashkelon
  - Ben Gurion University, Beersheba
  - Hadasit Medical Research Services & Development Ltd., Jerusalem
  - Rabin Medical Center, Petah Tikva
- Azienda Ospedaliera "Santi Antonio e Biagio e Cesare Arrigo, Allessandria, Italy
- P. Stradina Clinical University Hospital, Riga, Latvia
- Netherlands (3):
  - VU Amsterdam, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - Zaandam Medisch Centrum, Zaandam
- Hospital Nra. Sra. de Sonsoles, Ávila, Spain
- United Kingdom (6):
  - Selly Oak Hospital, Birmingham
  - St. Peter's Hospital / St. George's, Chertsey
  - Russels Hall Hospital, Dudley
  - University of Hull, Hull
  - Good Hope, Sutton Coldfield
  - Swansea NHS Trust, Swansea

REFERENCES:
- [Background] Ellery S, Pakrashi T, Paul V, Sack S. Predicting mortality and rehospitalization in heart failure patients with home monitoring--the Home CARE pilot study. Clin Res Cardiol. 2006;95 Suppl 3:III29-35. doi: 10.1007/s00392-006-1306-6. PMID 16598601
- [Derived] Sack S, Wende CM, Nagele H, Katz A, Bauer WR, Barr CS, Malinowski K, Schwacke H, Leyva F, Proff J, Berdyshev S, Paul V. Potential value of automated daily screening of cardiac resynchronization therapy defibrillator diagnostics for prediction of major cardiovascular events: results from Home-CARE (Home Monitoring in Cardiac Resynchronization Therapy) study. Eur J Heart Fail. 2011 Sep;13(9):1019-27. doi: 10.1093/eurjhf/hfr089. PMID 21852311